CLINICAL TRIAL: NCT02873338
Title: A Randomized, Phase II Study of CX-01 Combined With Standard Induction Therapy for Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Dociparstat Sodium (CX-01) Combined With Standard Induction Therapy for Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNTX-CX-01-2015-AML-1
Record Dates: First submitted 2016-08-12; First posted 2016-08-19 (Estimated); Results first posted 2021-10-29 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — N-desulfated,2-O,3-O-desulfated heparin; Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (idarubicin+cytarabine) (Active Comparator): Induction:
  * Idarubicin 12 mg/m2/day by slow (10 to 30 minutes) intravenous (IV) injection/infusion daily (Days 1, 2, and 3)
  * Cytarabine 100 mg/m2/day continuous 24-hour IV infusion (Days 1 to 7)
  Re-induction:
  * Idarubicin 12 mg/m2/day slow (10 to 30 minutes) IV injection/infusion daily (Days 1 and 2)
  * Cytarabine 100 mg/m2/day continuous 24-hour IV infusion (Days 1 to 5)
  Consolidation:
  • Cytarabine 1.0 g/m2 over 3 hours, every 12 hours (Days 1, 3, and 5)
  Interventions: Drug: Idarubicin; Drug: Cytarabine
- Dociparstat 0.125 mg/kg (Experimental): Induction:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-idarubicin dose (Day 1), followed by dociparstat 0.125 mg/kg/hr continuous 24-hour intravenous (IV) infusion (Days 1 to 7)
  * Idarubicin 12 mg/m2/day slow IV injection/infusion daily (Days 1, 2, and 3)
  * Cytarabine 100 mg/m2/day continuous 24-hour IV infusion (Days 1 to 7)
  Re-induction:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-idarubicin dose (Day 1), followed by dociparstat 0.125 mg/kg/hr continuous 24-hour IV infusion (Days 1 to 5)
  * Idarubicin 12 mg/m2/day slow IV injection/infusion daily (Days 1 and 2)
  * Cytarabine 100 mg/m2/day continuous 24-hour IV infusion (Days 1 to 5)
  Consolidation:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-3-hour cytarabine infusion (Day 1), followed by dociparstat 0.125 mg/kg/hr continuous 24-hour IV infusion on (Days 1 to 5; total 120 hours)
  * Cytarabine 1.0 g/m2 over 3 hours, every 12 hours (Days 1, 3, and 5)
  Interventions: Drug: Dociparstat sodium; Drug: Idarubicin; Drug: Cytarabine
- Dociparstat 0.25 mg/kg (Experimental): Induction:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-idarubicin dose (Day 1), followed by dociparstat 0.25 mg/kg/hr continuous 24-hour intravenous (IV) infusion (Days 1 to 7)
  * Idarubicin 12 mg/m2/day slow IV injection/infusion daily (Days 1, 2, and 3)
  * Cytarabine 100 mg/m2/day continuous 24-hour IV infusion (Days 1 to 7)
  Re-induction:
  * Dociparstat 4 mg/kg initial bolus 20 minutes post-idarubicin dose (Day 1), followed by dociparstat 0.25 mg/kg/hr continuous 24-hour IV infusion (Days 1 to 5)
  * Idarubicin 12 mg/m2/day slow IV injection/infusion daily (Days 1 and 2)
  * Cytarabine 100 mg/m2/day continuous 24-hour IV infusion (Days 1 to 5)
  Consolidation:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-3-hour cytarabine infusion (Day 1), followed by dociparstat 0.25 mg/kg/hr continuous 24-hour IV infusion (Days 1 to 5; total 120 hours)
  * Cytarabine 1.0 g/m2 over 3 hours, every 12 hours (Days 1, 3, and 5)
  Interventions: Drug: Dociparstat sodium; Drug: Idarubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: Dociparstat sodium — Subjects received 4 mg/kg dociparstat intravenous (IV) bolus followed by doses of 0.125 or 0.25 mg/kg/hr dociparstat given on Days 1 through 7 with standard induction therapy, on Days 1 through 5 or 7 with standard re-induction therapy, and on Days 1, 3, and 5 with standard consolidation therapy.
  Other Names: 2-O, 3-O desulfated heparin; ODSH; PGX-100; CX-01; Dociparstat
  Arms: Dociparstat 0.125 mg/kg; Dociparstat 0.25 mg/kg
Drug: Idarubicin — Subjects received 12 mg/m2/day idarubicin by slow (10 to 15 minutes) intravenous (IV) injection daily on Days 1, 2 and 3 of induction therapy, and on Days 1 and 2 of re-induction therapy.
  Other Names: Idamycin
Drug: Cytarabine — Subjects received 100 mg/m2/day cytarabine by continuous intravenous (IV) infusion on Days 1 through 7 of induction therapy and on Days 1 through 5 of re-induction therapy. During consolidation therapy, subjected received 1.0 g/m2 cytarabine IV infusion given over 3 hours every 12 hours on Days 1, 3, and 5.

SUMMARY:
This was an exploratory Phase 2, open label, randomized, multicenter, parallel group study to determine whether there was evidence that the addition of dociparstat (CX-01) at 2 different does levels to standard induction therapy (cytarabine+idarubicin, "7+3") and consolidation therapy had an additive therapeutic effect for subjects newly diagnosed with acute myeloid leukemia (AML) when compared with subjects receiving standard induction chemotherapy alone.

DETAILED DESCRIPTION:
The primary efficacy endpoint was to assess whether dociparstat in conjunction with standard induction therapy for AML increased the complete remission rate based on the International Working Group AML response criteria.

A total of 75 subjects were to be randomized in a 1:1:1 ratio to 1 of the following treatment groups:

* Group 1: cytarabine + idarubicin
* Group 2: cytarabine + idarubicin + dociparstat 0.125 mg/kg/hr
* Group 3: cytarabine + idarubicin + dociparstat 0.25 mg/kg/hr

Subjects received up to 2 induction cycles and up to 2 consolidation cycles and participated in the study for up to 18 months. Clinical laboratory tests were conducted routinely, and bone marrow aspirates and biopsies were performed during the induction cycles. Safety was monitored through adverse events and clinical laboratory results.

ELIGIBILITY:
Inclusion Criteria:

Subjects had to meet all the following criteria to be eligible for enrollment in this study:

1. Had newly diagnosed, de novo or secondary, previously untreated acute myeloid leukemia (AML).
2. Had an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.

Exclusion Criteria:

Subjects who met any of the following criteria were not eligible for enrollment in this study:

1. Had acute promyelocytic leukemia
2. Had prior chemotherapy for AML.
3. Had prior intensive chemotherapy or stem cell transplantation for the treatment of myelodysplastic syndrome.
4. Had central nervous system (CNS) leukemia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Marcus, MD, Study Director — Cantex Pharmaceuticals Inc.
Locations (23):
- United States (23):
  - University of California, San Diego, Moores Cancer Center, La Jolla, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - June E. Nylen Cancer Center, Sioux City, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Tulane University/Tulane Cancer Center, New Orleans, Louisiana
  - Karmanos Cancer Institute, Detroit, Michigan
  - Allina Health - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Northwell Health, Monter Cancer Center, Lake Success, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health & Science University Knight Cancer Institute, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Tennessee Oncology/Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor Research Institute/Baylor Sammons Cancer Center/Baylor University Medical Center, Dallas, Texas
  - Methodist Healthcare System of San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note that 2 randomized subjects did not receive study treatment: 1 subject in the control group and 1 subject in the dociparstat 0.25 mg/kg group. Therefore, these 2 subjects are not included in the safety analysis, but are included in the efficacy analyses.
Groups:
- Control (Idarubicin+Cytarabine): Induction:
  * Idarubicin 12 mg/m2/day by slow (10 to 30 minutes) intravenous (IV) injection/infusion daily (Days 1, 2, 3)
  * Cytarabine 100 mg/m2/day continuous 24-hr IV infusion (Days 1-7)
  Reinduction:
  * Idarubicin 12 mg/m2/day slow (10 to 30 minutes) IV injection/infusion daily (Days 1, 2)
  * Cytarabine 100 mg/m2/day continuous 24-hour IV infusion (Days 1-5)
  Consolidation:
  • Cytarabine 1.0 g/m2 over 3 hours, every 12 hours (Days 1, 3, 5)
- Dociparstat 0.125 mg/kg: Induction:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-idarubicin dose (Day 1), followed by dociparstat 0.125 mg/kg/h continuous 24-hr IV infusion (Days 1-7)
  * Idarubicin 12 mg/m2/day slow IV injection/infusion daily (Days 1, 2, 3)
  * Cytarabine 100 mg/m2/day continuous 24-hr IV infusion (Days 1-7)
  Reinduction:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-idarubicin dose (Day 1), followed by dociparstat 0.125 mg/kg/h continuous 24-hr IV infusion (Days 1-5)
  * Idarubicin 12 mg/m2/day slow IV injection/infusion daily (Days 1, 2)
  * Cytarabine 100 mg/m2/day continuous 24-hr IV infusion (Days 1-5)
  Consolidation:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-3-hour cytarabine infusion (Day 1), followed by dociparstat 0.125 mg/kg/h continuous 24-hr IV infusion on (Days 1-5; total 120 hours)
  * Cytarabine 1.0 g/m2 over 3 hrs, every 12 hrs (Days 1, 3, 5)
- Dociparstat 0.25 mg/kg: Induction:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-idarubicin dose (Day 1), followed by dociparstat 0.25 mg/kg/h continuous 24-hr IV infusion (Days 1-7)
  * Idarubicin 12 mg/m2/day slow IV injection/infusion daily (Days 1, 2, 3)
  * Cytarabine 100 mg/m2/day continuous 24-hr IV infusion (Days 1-7)
  Reinduction:
  * Dociparstat 4 mg/kg initial bolus 20 minutes post-idarubicin dose (Day 1), followed by dociparstat 0.25 mg/kg/h continuous 24-hr IV infusion (Days 1-5)
  * Idarubicin 12 mg/m2/day slow IV injection/infusion daily (Days 1, 2)
  * Cytarabine 100 mg/m2/day continuous 24-hr IV infusion (Days 1-5)
  Consolidation:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-3-hour cytarabine infusion (Day 1), followed by dociparstat 0.25 mg/kg/h continuous 24-hr IV infusion (Days 1-5; total 120 hours)
  * Cytarabine 1.0 g/m2 over 3 hours, every 12 hours (Days 1, 3, 5)
Period: Overall Study
Arm/Group | Control (Idarubicin+Cytarabine) | Dociparstat 0.125 mg/kg | Dociparstat 0.25 mg/kg
Started | 26 | 25 | 24
Completed | 8 | 4 | 6
Not Completed | 18 | 21 | 18
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Death | 2 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 3
Not completed — Lack of Efficacy | 0 | 2 | 0
Not completed — Other or Missing | 14 | 15 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Idarubicin+Cytarabine) | Dociparstat 0.125 mg/kg | Dociparstat 0.25 mg/kg | Total
Number analyzed (Participants) | 26 | 25 | 24 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (3.6) | 67 (4.8) | 68 (4.3) | 67 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 13 | 29
  Male | 20 | 15 | 11 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 4
  White | 23 | 22 | 20 | 65
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 3
Acute myeloid leukemia (AML) subtype [Count of Participants; unit: Participants]
  De novo | 22 | 18 | 22 | 62
  Secondary | 4 | 7 | 2 | 13
Time since acute myeloid leukemia (AML) diagnosis [Mean (Standard Deviation); unit: weeks] | 1.1 (1.19) | 1.2 (1.15) | 1.0 (0.75) | 1.1 (1.04)
Baseline blasts in bone marrow [Mean (Standard Deviation); unit: percentage] | 44 (25.9) | 47 (22.3) | 46 (26.6) | 46 (24.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Achieved Morphologic Complete Remission
Description: Morphologic complete remission (CR) was evaluated by International Working Group (IWG) criteria and defined as absolute neutrophil count (ANC) >1000/microliter; platelet count >100,000, <5% blasts in bone marrow aspirate, no blasts with Auer rods, and no evidence of extramedullary disease.
Time Frame: During induction and re-induction phases of treatment (up to 60 days after the start of each treatment cycle)
Measure: Count of Participants; unit: Participants
Groups:
- Dociparstat 0.125 mg/kg: Induction:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-idarubicin dose (Day 1), followed by dociparstat 0.125 mg/kg/hr continuous 24-hour intravenous (IV) infusion (Days 1 to 7)
  * Idarubicin 12 mg/m2/day slow IV injection/infusion daily (Days 1, 2, and 3)
  * Cytarabine 100 mg/m2/day continuous 24-hour IV infusion (Days 1 to 7)
  Re-induction:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-idarubicin dose (Day 1), followed by dociparstat 0.125 mg/kg/hr continuous 24-hour IV infusion (Days 1 to 5)
  * Idarubicin 12 mg/m2/day slow IV injection/infusion daily (Days 1 and 2)
  * Cytarabine 100 mg/m2/day continuous 24-hour IV infusion (Days 1 to 5)
  Consolidation:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-3-hour cytarabine infusion (Day 1), followed by dociparstat 0.125 mg/kg/h continuous 24-hour IV infusion on (Days 1 to 5; total 120 hours)
  * Cytarabine 1.0 g/m2 over 3 hours, every 12 hours (Days 1, 3, and 5)
Arm/Group | Control (Idarubicin+Cytarabine) | Dociparstat 0.125 mg/kg | Dociparstat 0.25 mg/kg
Number analyzed (Participants) | 26 | 25 | 24
Participants | 14 | 8 | 11

2. Secondary Outcome: Duration of Event-free Survival
Description: Event-free survival was measured as date of randomization until treatment failure. Treatment failure was defined as failure to achieve composite completed morphological remission during the induction and re-induction phase of the study lasting up to 60 days, relapse from complete response, or death from any cause, whichever occurred first.
Time Frame: Randomization up to 30 months
Population: Note: In the Dociparstat 0.125 mg/kg group, fewer than half of the subjects achieved complete CR, and thus were assessed as having an event on Day 1.
Measure: Median (Full Range); unit: days
Groups:
- Dociparstat 0.125 mg/kg: Induction:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-idarubicin dose (Day 1), followed by dociparstat 0.125 mg/kg/hr continuous 24-hour intravenous (IV) infusion (Days 1 to 7)
  * Idarubicin 12 mg/m2/day slow IV injection/infusion daily (Days 1, 2, and 3)
  * Cytarabine 100 mg/m2/day continuous 24-hour IV infusion (Days 1 to 7)
  Re-induction:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-idarubicin dose (Day 1), followed by dociparstat 0.125 mg/kg/hr continuous 24-hr IV infusion (Days 1 to 5)
  * Idarubicin 12 mg/m2/day slow IV injection/infusion daily (Days 1 and 2)
  * Cytarabine 100 mg/m2/day continuous 24-hour IV infusion (Days 1 to 5)
  Consolidation:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-3-hour cytarabine infusion (Day 1), followed by dociparstat 0.125 mg/kg/hr continuous 24-hr IV infusion on (Days 1 to 5; total 120 hours)
  * Cytarabine 1.0 g/m2 over 3 hours, every 12 hours (Days 1, 3, and 5)
- Dociparstat 0.25 mg/kg: Induction:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-idarubicin dose (Day 1), followed by dociparstat 0.25 mg/kg/hr continuous 24-hour intravenous (IV) infusion (Days 1 to 7)
  * Idarubicin 12 mg/m2/day slow IV injection/infusion daily (Days 1, 2, and 3)
  * Cytarabine 100 mg/m2/day continuous 24-hour IV infusion (Days 1 to 7)
  Re-induction:
  * Dociparstat 4 mg/kg initial bolus 20 minutes post-idarubicin dose (Day 1), followed by dociparstat 0.25 mg/kg/hr continuous 24-hr IV infusion (Days 1 to 5)
  * Idarubicin 12 mg/m2/day slow IV injection/infusion daily (Days 1 and 2)
  * Cytarabine 100 mg/m2/day continuous 24-hour IV infusion (Days 1 to 5)
  Consolidation:
  * Dociparstat 4 mg/kg initial bolus 30 minutes post-3-hour cytarabine infusion (Day 1), followed by dociparstat 0.25 mg/kg/hr continuous 24-hour IV infusion (Days 1 to 5; total 120 hours)
  * Cytarabine 1.0 g/m2 over 3 hours, every 12 hours (Days 1, 3, and 5)
Arm/Group | Control (Idarubicin+Cytarabine) | Dociparstat 0.125 mg/kg | Dociparstat 0.25 mg/kg
Number analyzed (Participants) | 26 | 25 | 24
days | 243.5 [1 to 853] | 1 [1 to 922] | 171.5 [1 to 842]

3. Secondary Outcome: Time to Leukemia-free Survival
Description: Leukemia-free survival was assessed as a secondary endpoint only in subjects who achieved composite complete remission and was measured from randomization until disease relapse or death from any cause, whichever occurred first. Assessments were performed every 3 months until death or 18 months after the last subject was randomized, whichever occurred first.
Time Frame: Randomization until disease relapse or patient death from any cause, whichever occurs first, assessed up to 30 months
Population: This analysis only included subjects who achieved composite complete remission. The following number of subjects were censored in each treatment group:
  * Control: 6/16 (37.5%) subjects
  * Dociparstat 0.125 mg/kg: 4/9 (44.4%) subjects
  * Dociparstat 0.25 mg/kg: 10/15 (66.7%) subjects
Measure: Median (Full Range); unit: days
Arm/Group | Control (Idarubicin+Cytarabine) | Dociparstat 0.125 mg/kg | Dociparstat 0.25 mg/kg
Number analyzed (Participants) | 16 | 9 | 15
days | 292 [1 to 581] | 448 [26 to 494] | 166 [1 to 315]

4. Secondary Outcome: Number of Subjects Who Achieved Overall Survival
Description: Overall survival was measured from the date of randomization until death from any cause. Assessments were performed every 3 months and continued until death or 18 months after the last patient was randomized, whichever came first.
Time Frame: Randomization to end of study (18 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Idarubicin+Cytarabine) | Dociparstat 0.125 mg/kg | Dociparstat 0.25 mg/kg
Number analyzed (Participants) | 26 | 25 | 24
Participants
  Subjects died | 14 | 14 | 9
  Subjects still alive | 12 | 11 | 15

5. Secondary Outcome: Number of Subjects Who Achieved Composite Complete Remission
Description: The composite complete remission (CR) rate included CR, CR without recovery of platelets (CRp), and CR without recovery of neutrophils and/or platelets (CRi), as defined by the International Working Group criteria during the induction and re-induction phases of treatment. CR was defined as an Absolute Neutrophil Count (ANC) >1000/μL, platelet count >100,000/μL, <5% blasts in bone marrow aspirate, no blasts with Auer rods, and no evidence of extramedullary disease. CRi was defined as an ANC <1000/μL and/or platelet count <100,000/, <5% blasts in bone marrow aspirate, no blasts with Auer rods, and no evidence of extramedullary disease.
Time Frame: Up to 60 days after the start of each treatment cycle
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Idarubicin+Cytarabine) | Dociparstat 0.125 mg/kg | Dociparstat 0.25 mg/kg
Number analyzed (Participants) | 26 | 25 | 24
Participants | 16 | 9 | 15

6. Secondary Outcome: Duration of Morphologic Complete Remission
Description: The duration of morphologic complete remission was assessed only in subjects who had achieved morphologic complete remission and was defined as the time from achievement of complete response to the detection or relapse. Relapse was defined as the reappearance of leukemia blasts in the peripheral blood, >5% blasts in the bone marrow not attributable to another cause, or appearance/reappearance of extramedullary disease and with a bone marrow blast percentage of >5% but ≤20%. If the latter, a repeat bone marrow examination was performed at least 7 days after the first marrow examination; documentation of the bone marrow blast percentage of >5% was necessary to establish relapse. Assessments were performed every 3 months and continued until death or 18 months after the last subject was randomized, whichever occurred first.
  Duration of morphologic complete remission (time from the achievement of complete response to the detection of relapse)
Time Frame: Randomization to end of study (18 months)
Population: This analysis only included subjects who had achieved morphologic complete remission.
  The following number of subjects were censored in each treatment group for this analysis; however the full ranges include censored subjects:
  * Control: 7/14 (50%) subjects
  * Dociparstat 0.125 mg/kg: 6/8 (75.0%) subjects
  * Dociparstat 0.25 mg/kg: 9/11 (81.8%) subjects
Measure: Median (Full Range); unit: days
Arm/Group | Control (Idarubicin+Cytarabine) | Dociparstat 0.125 mg/kg | Dociparstat 0.25 mg/kg
Number analyzed (Participants) | 14 | 8 | 11
days | 233 [1 to 451] | 494 [1 to 494] | 294 [1 to 315]

7. Secondary Outcome: Time to Recovery of Neutrophils
Description: Neutrophil recovery was assessed from randomization to Absolute Neutrophil Count (ANC) recovery (ANC >500/µL and >1000/µL) for up to 60 days after the start of each treatment cycle.
Time Frame: Randomization to ANC recovery, for up to 60 days after the start of each treatment cycle
Population: The following number of subjects were censored in each treatment group for both analyses (neutrophil recovery to >500/µL and >1000/µL):
  * Control: 6/26 (23.1%) subjects for both analyses (>500/µL and >1000/µL)
  * Dociparstat 0.125 mg/kg: 9/25 (36.0%) subjects for both analyses (>500/µL and >1000/µL)
  * Dociparstat 0.25 mg/kg: 7/24 (29.2%) subjects for >500/µL and 11/24 (45.8%) subjects for >1000/µL
Measure: Median (Full Range); unit: days
Arm/Group | Control (Idarubicin+Cytarabine) | Dociparstat 0.125 mg/kg | Dociparstat 0.25 mg/kg
Number analyzed (Participants) | 26 | 25 | 24
days
  Recovery to >500/µL: number analyzed (Participants) | 20 | 16 | 17
  Recovery to >500/µL | 32 [1 to 57] | 43 [9 to 70] | 29 [1 to 51]
  Recovery to >1000/µL: number analyzed (Participants) | 20 | 16 | 13
  Recovery to >1000/µL | 37 [1 to 64] | 42 [9 to 70] | 35 [1 to 57]

8. Secondary Outcome: Time to Platelet Recovery
Description: Platelet recovery was measured from randomization to platelet recovery (platelet count >20,000/µL and >100,000/µL)
Time Frame: Randomization to platelet recovery, for up to 60 days after the start of each treatment cycle
Population: The following number of subjects were censored in each treatment group for each analysis (platelet recovery to >20,000µL and >100,000µL):
  * Control: 5/26 (19.2%) subjects for >20,000µL and 7/26 (26.9%) subjects for >100,000µL
  * Dociparstat 0.125 mg/kg: 5/25 (20%) subjects for >20,000µL and 12/25 (48.0%) subjects for >100,000µL
  * Dociparstat 0.25 mg/kg: 8/24 (33.3%) subjects for >20,000µL and 11/24 (45.8%) subjects for >100,000µL
Measure: Median (Full Range); unit: days
Arm/Group | Control (Idarubicin+Cytarabine) | Dociparstat 0.125 mg/kg | Dociparstat 0.25 mg/kg
Number analyzed (Participants) | 26 | 25 | 24
days
  Recovery to >20,000µL: number analyzed (Participants) | 21 | 20 | 16
  Recovery to >20,000µL | 35 [1 to 71] | 36 [16 to 70] | 29 [1 to 56]
  Recovery to >100,000µL: number analyzed (Participants) | 19 | 13 | 13
  Recovery to >100,000µL | 38 [1 to 71] | 50 [16 to 70] | 32 [1 to 56]

9. Secondary Outcome: Number of Subjects Who Died by Day 30
Description: Mortality (rate of death) of subjects by Day 30, measured from the first day of induction treatment to 30 days post-induction.
Time Frame: 30 days (from first day of induction treatment to 30 days after)
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Idarubicin+Cytarabine) | Dociparstat 0.125 mg/kg | Dociparstat 0.25 mg/kg
Number analyzed (Participants) | 26 | 25 | 24
Participants | 2 | 1 | 3

10. Secondary Outcome: Number of Subjects Who Died by Day 60.
Description: Mortality (rate of death) of subjects by Day 60, measured from the first day of induction treatment to 60 days post-induction.
Time Frame: 60 days (from the first day of induction treatment to 60 days after)
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Idarubicin+Cytarabine) | Dociparstat 0.125 mg/kg | Dociparstat 0.25 mg/kg
Number analyzed (Participants) | 26 | 25 | 24
Participants | 2 | 2 | 3

11. Secondary Outcome: Number of Subjects Who Died by Day 90
Description: Mortality (rate of death) of subjects at Day 90, measured from the first day of induction treatment to 90 days post-induction.
Time Frame: 90 days (from the first day of induction treatment to 90 days after)
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Idarubicin+Cytarabine) | Dociparstat 0.125 mg/kg | Dociparstat 0.25 mg/kg
Number analyzed (Participants) | 26 | 25 | 24
Participants | 2 | 3 | 3

ADVERSE EVENTS:
Time Frame: From signing informed consent to end of study (up to 30 months)
Description: Note that all-cause mortality was assessed for all randomized participants and adverse events were monitored for only participants who received at least 1 dose of study drug; 2 participants (1 in the control group and 1 in the 0.25 mg/kg dociparstat group) were randomized but did not receive study drug and were therefore not monitored for adverse events.
Arm/Group | Control (Idarubicin+Cytarabine) | Dociparstat 0.125 mg/kg | Dociparstat 0.25 mg/kg
All-Cause Mortality (participants affected / at risk) | 14/26 | 14/25 | 9/24
Serious Adverse Events (participants affected / at risk) | 7/25 | 8/25 | 13/23
Other Adverse Events (participants affected / at risk) | 25/25 | 25/25 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (Idarubicin+Cytarabine) (N=25) | Dociparstat 0.125 mg/kg (N=25) | Dociparstat 0.25 mg/kg (N=23)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (Idarubicin+Cytarabine) (N=25) | Dociparstat 0.125 mg/kg (N=25) | Dociparstat 0.25 mg/kg (N=23)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 16 | 17
Anaemia (Blood and lymphatic system disorders) | 13 | 12 | 8
Neutropenia (Blood and lymphatic system disorders) | 6 | 5 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 4 | 3
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 3 | 1
Tachycardia (Cardiac disorders) | 1 | 3 | 0
Atrial flutter (Cardiac disorders) | 2 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0
Vision blurred (Eye disorders) | 1 | 2 | 1
Eye irritation (Eye disorders) | 2 | 1 | 0
Eye pain (Eye disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 16 | 15 | 15
Diarrhoea (Gastrointestinal disorders) | 14 | 14 | 15
Constipation (Gastrointestinal disorders) | 10 | 7 | 9
Abdominal pain (Gastrointestinal disorders) | 8 | 5 | 9
Vomiting (Gastrointestinal disorders) | 6 | 4 | 8
Stomatitis (Gastrointestinal disorders) | 4 | 6 | 5
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 7
Flatulence (Gastrointestinal disorders) | 2 | 6 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 4 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 5 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 6 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2
Chapped lips (Gastrointestinal disorders) | 2 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 2 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 3 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 2 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 2 | 1
Gingival pain (Gastrointestinal disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 14 | 16 | 12
Pyrexia (General disorders) | 13 | 8 | 9
Fatigue (General disorders) | 6 | 11 | 10
Chills (General disorders) | 6 | 5 | 4
Mucosal inflammation (General disorders) | 1 | 4 | 4
Peripheral swelling (General disorders) | 1 | 2 | 2
Localised oedema (General disorders) | 2 | 1 | 0
Oedema (General disorders) | 1 | 0 | 2
Injection site bruising (General disorders) | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 2 | 3
Sepsis (Infections and infestations) | 2 | 3 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 3 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 2
Candida infection (Infections and infestations) | 0 | 1 | 2
Enterococcal infection (Infections and infestations) | 1 | 2 | 0
Pneumonia fungal (Infections and infestations) | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 2 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 3 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Platelet count decreased (Investigations) | 8 | 9 | 7
White blood cell count decreased (Investigations) | 6 | 7 | 7
Aspartate aminotransferase increased (Investigations) | 5 | 5 | 5
Neutrophil count decreased (Investigations) | 4 | 4 | 7
Alanine aminotransferase increased (Investigations) | 4 | 6 | 4
Lymphocyte count decreased (Investigations) | 2 | 4 | 6
Blood bilirubin increased (Investigations) | 1 | 4 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 2 | 3
Blood creatinine increased (Investigations) | 2 | 1 | 1
Weight decreased (Investigations) | 1 | 1 | 2
International normalised ration increased (Investigations) | 0 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 16 | 13
Decreased appetite (Metabolism and nutrition disorders) | 7 | 10 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 9 | 8 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 5 | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 6 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 4 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 7 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3 | 3
Fluid overload (Metabolism and nutrition disorders) | 1 | 4 | 1
Alkalosis (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 2 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 3 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 6 | 9 | 6
Dizziness (Nervous system disorders) | 5 | 5 | 4
Dysgeusia (Nervous system disorders) | 1 | 2 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 2
Syncope (Nervous system disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 8 | 6 | 6
Anxiety (Psychiatric disorders) | 4 | 2 | 3
Confusional state (Psychiatric disorders) | 0 | 3 | 3
Depression (Psychiatric disorders) | 1 | 0 | 5
Hallucination (Psychiatric disorders) | 1 | 4 | 1
Delirium (Psychiatric disorders) | 3 | 1 | 1
Agitation (Psychiatric disorders) | 1 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 4 | 1 | 4
Acute kidney injury (Renal and urinary disorders) | 1 | 3 | 2
Haematuria (Renal and urinary disorders) | 2 | 2 | 2
Dysuria (Renal and urinary disorders) | 0 | 3 | 2
Urinary retention (Renal and urinary disorders) | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 7 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 4 | 6 | 6
Hypotension (Vascular disorders) | 4 | 4 | 3
Deep vein thrombosis (Vascular disorders) | 2 | 4 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the Study and its results shall not be publicized or published in any form without prior consent of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-01-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT02873338/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT02873338/SAP_001.pdf